CLINICAL TRIAL: NCT06908421
Title: A 52-week, Multicentre, Observational, Prospective Study on the Use of a Smart Platform Connected to a Single-inhaler Triple Therapy (ICS/LABA/LAMA) to Evaluate Effectiveness on Treatment Adherence and Inhaler Technique in Patients With Poorly Controlled Asthma.
Brief Title: Efficacy of a Smart add-on Device in Combination With a Triple Treatment in Asthma Patients on Inhaler Technique and Adherence
Acronym: SiASMARTer
Status: Recruiting | Type: Observational
Sponsor: Chiesi Pharma AB, Nordic (Industry)
Collaborators: Briota ApS (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-193-23
Record Dates: First submitted 2025-03-17; First posted 2025-04-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Asthma; Inhaler treatment; smart add-on device; adherence; inhaler technique
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: Asthma patients above 18 years of age, with objectively verified diagnosis of asthma according to GINA, uncontrolled T2 inflammation (FeNO >25ppm) on BDP/FF/G inhalation treatment with prescribed rescue medication (SABA).

SUMMARY:
The goal of this observational study is to determine if using the SiA® (Systematic Intervention Agent) system can improve inhaler technique and medication adherence in adults with asthma who are already using Trimbow pMDI inhalers. Furthermore, it will be addressed if the SiA® system can be used to discriminate between patients, where increased inflammatory markers are caused by incorrect inhaler technique/adherence to medication or patients that have ongoing inflammation requiring adjustment of therapy. Potentially those who might become candidate for biological treatments.

The main questions it aims to answer are:

* Can the SiA® system improve inhaler use and medication adherence in asthma patients?
* Does improving inhaler technique and adherence lead to better asthma control and reduced airway inflammation (measured by FeNO levels)?

Participants will:

* Use the SiA® system, which includes a smart inhaler cap (RespiPRO™) and a mobile app
* Continue their prescribed Trimbow pMDI treatment for asthma.
* Have their asthma control, lung function, and FeNO levels monitored at specific points over 1 year (3 months and 12 months).

The study does not have a comparison group and all results will be compared to baseline.

DETAILED DESCRIPTION:
Background and Rationale Asthma is a chronic inflammatory disease of the airways that affects millions of individuals worldwide. Despite the availability of effective inhaled medications, poor adherence and incorrect inhaler technique remain major barriers to optimal asthma control. Studies show that up to 86.7% of asthma patients make at least one inhaler technique error, and 30-40% demonstrate poor adherence to their prescribed medication. These factors contribute to worsened symptoms, increased healthcare utilization, and reduced quality of life.

The SiA® system, developed by Briota ApS, aims to address these challenges by integrating a smart inhaler cap (RespiPRO™) with a mobile application. This system provides real-time feedback on inhaler technique and adherence, allowing patients and healthcare providers to track progress and make necessary adjustments.

This study seeks to determine whether using the SiA® system alongside a pressurized metered dose inhaler (pMDI) therapy can lead to measurable improvements in medication adherence, inhalation technique, and asthma control. Furthermore, it will be addressed if the SiA® system can be used to discriminate between patients, where increased inflammatory markers are caused by inadequate treatment caused by incorrect inhaler technique/adherence to medication or patients that have ongoing inflammation requiring adjustment of therapy. Potentially those who might become candidate for biological treatments.

Study Design This is a prospective, single-arm observational study conducted at two hospitals in Denmark. It is designed to assess how the SiA® System impacts inhaler technique and medication adherence over a 12-month period.

Key Features of the Study Design:

* Observational (non-interventional): Participants will continue their standard asthma medication (Trimbow pMDI) but will use the SiA® system to monitor their inhaler technique and adherence.
* Single-arm design: All participants will receive the SiA® System - there is no comparison group.
* Real-world setting: The study aims to reflect how patients interact with the SiA® system in everyday life, outside of a controlled clinical trial environment.

Study Setting:

* Conducted at two specialized respiratory clinics in Denmark.
* Participants will be recruited from routine asthma care visits.

Data Collection Methods:

Data will be collected through multiple sources:

* Hospital medical records (to gather historical asthma data and prior exacerbation history).
* Spirometry tests (to assess lung function).
* FeNO tests (to measure airway inflammation).
* SiA® System data (to track inhaler adherence and technique).
* Patient-reported outcome measures (questionnaires on asthma symptoms and quality of life).

Technology Used in the Study:

* RespiPRO™ Smart Inhaler Cap: A device that attaches to Trimbow pMDI and records inhaler usage data.
* SiA® Mobile App: Tracks daily inhaler use, provides feedback, and sends adherence reminders.

Study Timeline:

Total Study Duration: 22 months, with individual patient follow-up lasting 12 months (52 weeks).

Patient Flow and Study Visits:

1. Screening and Baseline Visit (Week 0) - Study Enrolment

   * Patients will be identified during routine asthma care visits and screened for eligibility.
   * Informed consent will be obtained.
   * Baseline data collection will include:
   * Medical history
   * Asthma severity and medication use
   * Spirometry test (lung function)
   * FeNO test (airway inflammation)
   * ACT (Asthma Control Test) and mini-AQLQ (Asthma Quality of Life Questionnaire)
   * Patients will receive a brief training session on how to use the SiA® System.
   * A baseline inhaler technique video will be recorded using the SiA® Mobile App.
2. Interim Follow-up Visit (Week 12) - Progress Check

   * Patients will return for an in-person visit.
   * Repeat measurements:

     * FeNO test (to check inflammation levels).
     * Spirometry (lung function test).
     * ACT and mini-AQLQ (patient-reported outcomes).
   * Adherence data from the SiA® system will be reviewed.
   * Patients will complete a satisfaction survey about their experience with the SiA® system.
3. Final Study Visit (Week 52) - End of Study

   * Repeat FeNO, spirometry, ACT, and mini-AQLQ assessments.
   * The final inhaler technique video will be recorded and analyzed.
   * Patients will return or deactivate the RespiPRO™ Smart Inhaler Cap.
   * Final adherence and inhalation technique data will be collected from the SiA® Dashboard.

Potential Impact of the Study

This study aims to generate real-world evidence on how digital health interventions can improve asthma management. If successful, the SiA® System could:

* Enhance asthma control by ensuring patients use their inhalers correctly.
* Reduce unnecessary medication escalation, preventing overuse of corticosteroids.
* Lower healthcare costs by reducing asthma-related hospital visits.
* Empower patients with real-time feedback and better self-management tools.
* Improve and optimize the way asthma patients become candidate for biological treatments

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age.
2. Objectively verified leading diagnosis of asthma according to GINA
3. FeNO >25 ppb.
4. Treated with Trimbow 87/5/9 pMDI for >4 weeks before enrolment,

   1. with prescribed rescue medication (SABA).
   2. with and without prescription of a spacer.
5. Being literate Danish.
6. Having a personal Android/iOS phone and 4G/5G internet connection.
7. Comfortable using a smart phone and Bluetooth enabled Digital Devices.
8. Willingness to participate in the study, understand the written patient information and being able to provide written informed consent.

Exclusion Criteria:

1. Participation in a clinical trial within 4 weeks prior to enrolment into the present study or planned enrolment in a clinical trial during the observational period.
2. Use of systemic corticosteroid as maintenance treatment.
3. Treated with biologics (that is monoclonal antibodies).
4. Concomitant diagnosis of COPD.
5. Lung cancer or history of lung cancer.
6. Respiratory tract infection/exacerbation within 4 weeks prior to enrolment.
7. Use of oral corticosteroids within 4 weeks before enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients above 18 years of age, with objectively verified diagnosis of asthma according to GINA, uncontrolled T2 inflammation (FeNO >25ppm) on BDP/FF/G inhalation treatment with prescribed rescue medication (SABA).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of the SiA® platform on the level of the type 2 inflammation biomarker FeNO | Change from baseline in FeNO at week 12 and 52.
  To assess the impact of the study on the type 2 biomarker FeNO with a change from baseline of at least 20% will be considered clinically relevant. FeNO values will be presented as ppb. FeNO levels of < 25 ppb, 25 - 50 ppb, > 50 ppb, are considered low, medium, and high respectively.

SECONDARY OUTCOMES:
To assess the impact of the SiA® platform on adherence to SITT and inhaler technique measure using the RespiPRO add-on module | Change in pMDI inhaler technique score and medication adherence score at week 12 and 52 compared to baseline.
  Change in inhaler adherence measured as percentage of days covered and inhaler technique scores based an assessments of inhalation video recordings an data collected from the SiA® platform using a scoring system of 1-5, where 5 = Optimal technique; 4 = Poor technique with one critical error; 3 = Poor technique with two critical errors; ≤2 = Poor technique with three or more critical errors. The RespiPRO™ cannot monitor step 1 and 2, thus are these by default set to 1, hence the minimum inhaler technique scores achievable from RespiPRO™ is 2.
To evaluate the impact of the SiA® platform on asthma control using Asthma Control Test | Change in ACT scores from baseline at weeks 12 and 52
  Asthma control will be assesed using Asthma Control Test (ACT), which is a patient self-administred tool for identifying those with poorly controlled asthma. A maximum score of 25 points indicates complete asthma control. A score between 20 and 25 represents well controlled asthma, while a score of 19 or below represents not well controlled asthma, and a score less than 16 indicates very poorly controlled asthma.
To evaluate the impact of the SiA® platform on health-related quality of life | Change in mini-AQLQ scores from baseline at weeks 12 and 52
  To assess the impact of the study on Health-related Quality of Life (HR QoL) using Asthma Quality of Life Questionnaire (mini-AQLQ). The mini-AQLQ has 15 questions in the same domains as the original AQLQ (symptoms, activities, emotions and environment).
To evaluate the impact of the SiA® platform on lung function measured by spirometry | From baseline and at week 12 and 52.
  Change in lung function parameters (change in mean FEV1, FEV1 %-predicted, FEV1/FVC ratio, FEF25-75) from baseline at weeks 12 and 52
To evaluate the impact of the SiA® platform on shifts in FeNO category | Change from baseline at week 12 and 52.
  Change in FeNO category (low, intermediate, high) defined as (< 25 ppb, 25 - 50 ppb, > 50 ppb, respectively.
To evaluate the impact of the SiA® platform on annualized exacerbations rates | Change in annualized exacerbation rates (moderate and severe) from baseline at week 52
  Retrospective data from the past 12 months will gathered the number of moderate and severe exacerbations as defined by the American Thoracic Society/European Respiratory Society.
o evaluate the impact of the SiA® platform on the use of rescue medication (SABA) | Change from baseline (first 7 days after entering the study) in the use of rescue medication (SABA) at week 12 and 52).
  To assess the impact of the study intervention on use of rescue medication (SABA) measured as average puffs per day/week/month.
Satisfaction and compliance with add-on device based on a customized survey | at week 52.
  Satisfaction score at week 52 assessed using a customized questionnaire. The survey reports on 9 question related to the satisfaction with SiA® platform. Each of the 9 question can be given a score from 1-5. where 1 = very difficult/dissatisfied, 3 = neutral, and 5 = very easy/satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes M Schmid, PhD, ass. professor, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital-Hvidovre, Hvidovre, Capital Region
  - Aarhus University Hospital, Aarhus, Central Jutland

IPD SHARING:
Plan to Share IPD: Undecided